CLINICAL TRIAL: NCT06060145
Title: Effect of Indoor Plants on Cardiopulmonary System: a Randomized, Crossover, Controlled Trial
Brief Title: Effect of Indoor Plants on Cardiopulmonary System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lina Zhang (Other Government)
Collaborators: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Sponsor-Investigator, Lina Zhang, Lecturer, Zhejiang Chinese Medical University
Organization: Zhejiang Chinese Medical University (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 20230922-4
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Cardiopulmonary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plants placed in an office environment (Experimental): Participants in this group will receive an intervention of plants placed in an office environment.
  Interventions: Other: Plants placed in an office environment
- Devoid of any plant presence in an office environment (Active Comparator): Participants in this group will be exposed to an office environment devoid of any plant presence.
  Interventions: Other: Devoid of any plant presence in an office environment

INTERVENTIONS:
Other: Plants placed in an office environment — The intervention group will be provided with an intervention consisting of 34-38 potted plants arranged in an office environment for a duration of 8 hours (09:00-17:00) on weekdays (Monday to Friday) for 4 weeks.
  Arms: Plants placed in an office environment
Other: Devoid of any plant presence in an office environment — Participants assigned to the control group will be exposed to an office environment devoid of any plant presence for a duration of 8 hours (09:00-17:00) on weekdays (Monday to Friday) for 4 weeks.
  Arms: Devoid of any plant presence in an office environment

SUMMARY:
This is a randomized controlled human exposure crossover study, aims to explore the health benefits of indoor plants on cardiopulmonary system on adults.

DETAILED DESCRIPTION:
The researchers will conduct a randomized cross-controlled trial involving 48 healthy adults in Hangzhou, China. These participants will be randomly assigned into two groups, each comprising 24 individuals. Each participant will undergo two separate exposures in an office setting: one exposure without any plants present, and another exposure with 34 to 38 potted plants. A washout period of at least 4 weeks will be implemented between the two exposures. Questionnaires, physical examinations and the collection of biological samples will be conducted prior to exposure and after exposure. In addition, the monitoring of negative air ion, air pollutants and noise exposure, as well as collection of environmental microbial samples, will be conducted on weekdays. Researchers will gather samples of blood, urine, nasal secretion, and exhaled breath condensate from participants.

ELIGIBILITY:
Inclusion Criteria:

* Living in Hangzhou during the study period;
* Non-smoking, no history of alcohol or drug abuse;
* Staying indoors in daytime we required.

Exclusion Criteria:

* Current or ever smokers;
* Subjects with allergic disease, such as allergic rhinitis, allergic asthma, and atopy;
* Subjects with cardiovascular disease, such as congenital heart disease, pulmonary heart disease, and hypertension;
* Subjects with respiratory disease, such as asthma, chronic bronchitis, and chronic obstructive pulmonary disease;
* Subjects with chronic disease, such as diabetes, chronic hepatitis, and kidney disease;
* Subjects with a history of major surgery;
* Medication use or dietary supplements intake in recent two months;
* Unable to cooperate with follow-up.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity(FVC) | Baseline and after 4 weeks plants exposure in first stage, and after washout period, baseline and after 4 weeks plants exposure in second stage.
  We plan to measure forced vital capacity (FVC) of lung function.

SECONDARY OUTCOMES:
Blood Pressure(BP) | Baseline and after 4 weeks plants exposure in first stage, and after washout period, baseline and after 4 weeks plants exposure in second stage.
  We plan to measure systolic blood pressure (SBP) and diastolic blood pressure (DBP).
Heart Rate Variability(HRV) | Baseline and after 4 weeks plants exposure in first stage, and after washout period, baseline and after 4 weeks plants exposure in second stage.
  We plan to measure Heart Rate Variability (HRV).

OTHER OUTCOMES:
C-reactive protein(CRP) | Baseline and after 4 weeks plants exposure in first stage, and after washout period, baseline and after 4 weeks plants exposure in second stage.
  We plan to measure serum concentrations of C-reactive protein(CRP)
Interleukin-6(IL-6) | Baseline and after 4 weeks plants exposure in first stage, and after washout period, baseline and after 4 weeks plants exposure in second stage.
  We plan to measure the serum concentrations of Interleukin-6
Tumor necrosis factor-α(TNF-α) | Time Frame: Baseline and after 4 weeks plants exposure in first stage, and after washout period, baseline and after 4 weeks plants exposure in second stage.
  We plan to measure the serum concentrations of Tumor necrosis factor-α

CONTACTS AND LOCATIONS:
Overall Officials: Lina Zhang, Ph.D, Principal Investigator — School of Public Health, Zhejiang Chinese Medical University
Locations (1):
- Zhejiang Chinese Medicine University, Huangzhou, Zhejiang, China